CLINICAL TRIAL: NCT02673710
Title: A Multicenter Non-Interventional Study Exploring the Impact of Sarcopenia on the Outcomes of Colorectal Cancer Patients Treated With a Chemotherapy Combined With Bevacizumab
Brief Title: A Study to Assess the Impact of Sarcopenia on the Outcomes of Colorectal Cancer Patients Treated With Chemotherapy Combined With Bevacizumab
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29985
Record Dates: First submitted 2016-01-27; First posted 2016-02-04 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Participants with metastatic colorectal cancer: Participants diagnosed with mCRC treated in first line with a combination of bevacizumab and chemotherapy for whom it is decided to continue the administration of bevacizumab beyond progression while changing CTR will be included in this study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Besides participant reported outcomes and a muscle strength test no interventions are administered, all treatment decisions are at the discretion of the physician and will be in line with local clinical practice and labeling

SUMMARY:
The purpose of this study is to explore the relationship between sarcopenia, as defined by computed tomography, treatment related outcomes and other body composition related parameters in a patient population receiving bevacizumab beyond progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in first line with bevacizumab for whom it is decided, and who are clinically considered eligible, to continue the treatment with bevacizumab beyond PD1.
* Women of childbearing potential have to use effective contraception during (and up to 6 months after) treatment.
* Availability of specific retrospective data at diagnosis and during 1st line treatment

Exclusion Criteria:

* Patients who are participating or participated in first line in any other interventional clinical trial involving non-standard of care procedures impacting the body composition
* Dementia or another mental condition making it impossible to fill out questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with mCRC treated in first line with a combination of bevacizumab and chemotherapy for whom it is decided to continue the administration of bevacizumab beyond progression while changing chemotherapy regimen (CTR) will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Second Progression Free Survival (PFS2) defined as the time interval between study entry and the date of progression or death for any cause, whichever occurs first | Up to 3 years
Sarcopenia quantified via CT-scan defined as a skeletal muscle index at the 3rd lumbar vertebra below 41 for women and below 43 or 53 for men with a Body Mass Index below or above 25 respectively | Up to 3 years

SECONDARY OUTCOMES:
Participants body weight at initial diagnosis of mCRC | Up to 3 years
Participants body mass index at initial diagnosis of mCRC | Up to 3 years
Participants skeletal muscle mass at initial diagnosis of mCRC | Up to 3 years
Participants visceral fat mass, subcutaneous fat mass, total fat mass at SE | Up to 3 years
Participants Eastern Cooperative Oncology Group Performance status at SE | Up to 3 years
Participant muscle strength at initial diagnosis of mCRC | Up to 3 years
Participants primary and metastases location at Initial Diagnosis | Up to 3 years
Participants mutation status at Initial Diagnosis | Up to 3 years
Participants C-Reactive Protein and Albumin blood values at Initial Diagnosis | Up to 3 years
Participants Date of diagnosis of non-metastatic CRC disease at Initial Diagnosis | Up to 3 years
Participant with 1st line Chemotherapeutic regimen at Initial Diagnosis | Up to 3 years
Functional status using Functional Assessment for Cancer Treatment - specific for Colorectal cancer participants | Up to 3 years
Participant Physical status expressed in muscle strength | Up to 3 years
Participant Physical status expressed in Body Weight | Up to 3 years
Participant Physical status expressed in Body Mass Index | Up to 3 years
Nutritional status using the Patient-Generated Subjective Global Assessment questionnaire | Up to 3 years
Nutritional status using Visual Analogue Scale for appetite | Up to 3 years
Treatment related toxicity using MD Anderson Symptom Inventory scale | Up to 3 years
Number of participants with Number of chemotherapy cycles | Up to 3 years
Number of participants with Number of bevacizumab administrations | Up to 3 years
Number of participants with Treatment changes and treatment (un)changed until Second Progressive Disease | Up to 3 years
Number of participants with Reason for treatment changes | Up to 3 years
Intake dietary supplements | Up to 3 years
Dietary and physical counselling | Up to 3 years
Number of Participants with Adverse Events | Up to 3 years
First Progression Free Survival (PFS1) is defined as the time between initial diagnosis and first progressive disease | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Belgium (23):
  - Onze Lieve Vrouwziekenhuis Aalst, Aalst
  - AZ Sint Lucas Brugge, Assebroek
  - CHIREC, Auderghem
  - Imeldaziekenhuis, Bonheiden
  - AZ KLINA, Brasschaat
  - AZ Sint Jan, Bruges
  - Institut Jules Bordet X, Brussels
  - Hospital Erasme, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - Grand Hôpital de Charleroi Notre Dame, Charleroi
  - AZ Maria Middelares, Ghent
  - Jessa Zkh (Campus Salvator), Hasselt
  - UZ Leuven Gasthuisberg, Leuven
  - CHC MontLégia, Liège
  - CHU Sart-Tilman, Liège
  - AZ St Maarten Campus Leopoldstr, Mechelen
  - Hôpital André Vésale, Montigny-le-Tilleul
  - AZ Damiaan, Ostend
  - AZ Delta (Campus Wilgenstraat), Roeselare
  - AZ Glorieux- vzw Werken Glorieux, Ronse
  - AZ Nikolaas (Sint Niklaas), Sint-Niklaas
  - AZ Turnhout Sint Elisabeth, Turnhout
  - CHR de Verviers - East Belgium, Verviers